CLINICAL TRIAL: NCT00511771
Title: A Treatment Investigational New Drug (tIND) Program of Tegaserod 6 mg Bid Given Orally in Women Adult Patients With Irritable Bowel Syndrome With Constipation or With Chronic Idiopathic Constipation
Brief Title: A Treatment Investigational New Drug (tIND) Program of Tegaserod in Women With Irritable Bowel Syndrome With Constipation or With Chronic Idiopathic Constipation
Status: No longer available | Type: Expanded Access
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Other Study IDs: CHTF919A2433
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Irritable Bowel Syndrome With Constipation; Chronic Idiopathic Constipation
Keywords: Tegaserod, treatment IND, irritable bowel syndrome with constipation, IBS-C, chronic idiopathic constipation, CIC, chronic constipation, CC
MeSH Terms: interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod — Tegaserod maleate
  Other Names: Zelnorm

SUMMARY:
To provide tegaserod to eligible women adult patients who did not have satisfactory improvement of their irritable bowel syndrome with constipation (IBS-C) or chronic idiopathic constipation (CIC) symptoms with other available treatment(s) and / or patients who had satisfactory improvement of their symptoms with prior tegaserod treatment for IBS-C or CIC.

ELIGIBILITY:
Inclusion Criteria:

1. For patients with IBS-C: Women of 18-54 years of age with IBS-C according to the Rome III criteria.
2. For patients with Chronic Idiopathic Constipation: Women of 18-54 years of age with CIC according to the Rome III criteria .
3. Patients who did not have satisfactory symptom improvement of their IBS-C or CIC symptoms with other available treatment(s) and / or patients who had satisfactory improvement of their symptoms with prior tegaserod treatment for IBS-C or CIC. Satisfactory symptom improvement will be assessed by the patient.
4. Patients signed the informed consent

Exclusion Criteria:

1. History of or current diagnosis of cardiovascular ischemic disease (e.g., angina pectoris, myocardial infarction, transient ischemic attack or stroke and including findings suggestive of ischemia on an ECG such as changes in ST segment and T waves, and / or Q wave)
2. Patients who have uninvestigated symptoms suggestive of a cardiovascular ischaemic disease such as chest pain or chest discomfort, shortness of breath, sudden onset of weakness of the arms or the legs, difficult talking or loss of sensation etc
3. Presence of any cardiovascular risk factors according to the NIH guideline [NIH Publication No. 01-3670] (such as hypertension, hyperlipidemia, diabetes mellitus, active smoking, obesity and family history of premature coronary heart disease) as assessed by the investigator
4. Clinical evidence of significant (as judged by the Investigator) respiratory, cardiovascular, renal, hepatic-biliary, endocrine, psychiatric or neurologic diseases or presence of abdominal adhesions
5. History of or current eating disorder such as anorexia or bulimia or compulsory overeating.
6. Uncompensated depression or anxiety or suicidal ideation or behavior.
7. Diagnosis of mega-rectum or colon, a history of intestinal obstruction, congenital anorectal malformation, clinically significant rectocele, or any evidence of intestinal structural abnormality including gastrointestinal resection that affected bowel transit or any evidence of intestinal carcinoma, of inflammatory bowel disease or of alarm symptoms such as weight loss, rectal bleeding, or anemia
8. Evidence of cathartic colon or a history of drug (including laxative) or alcohol abuse, that in the Investigator's opinion, the patient is likely to continue to abuse these substances during the tIND program period
9. Pregnant women or breastfeeding women; fertile women who are not currently practicing medically approved method of contraception
10. Participating in other investigational studies concurrently or within 1 month prior to entering this tIND program
11. Hypersensitive to tegaserod or to any of the excipients
12. Patients who had tolerability or safety concerns with prior use of tegaserod.

Ages: 18 Years to 54 Years | Sex: Female
Age Groups: Adult